CLINICAL TRIAL: NCT07293260
Title: A Double-blind, Randomized, Placebo-controlled, Multi-center Study Evaluating the Safety, Tolerability, and Effect of Olpasiran on Coronary Artery Plaque Burden Assessed by Coronary Computed Tomography Angiography in Participants With Stable Atherosclerotic Cardiovascular Disease and Elevated Lipoprotein(a)
Brief Title: Olpasiran Trials of Cardiovascular Events and Lipoprotein(a) Reduction - Coronary Computed Tomography Angiography Trial
Acronym: OCEAN(a)-CCTA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230191
Expanded Access: NCT07079267 (Available)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Disease
Keywords: Stable Atherosclerotic Cardiovascular Disease; Elevated Lipoprotein(a); Coronary Artery Plaque Burden; Olpasiran
MeSH Terms: conditions — Cardiovascular Diseases | interventions — olpasiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olpasiran (Experimental): Participants will receive olpasiran subcutaneously (SC) once every 12 weeks (Q12W).
  Interventions: Drug: Olpasiran
- Placebo (Placebo Comparator): Participants will receive placebo SC Q12W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olpasiran — Olpasiran will be administered SC.
  Other Names: AMG 890
  Arms: Olpasiran
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to evaluate the effect of olpasiran, compared to placebo, on non-calcified plaque (NCP) volume as measured by Coronary Computed Tomography Angiography (CCTA).

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to ≤ 80 years.
* Lp(a) ≥ 200 nmol/L during screening.
* Angiographic evidence of coronary artery disease in at least one major epicardial vessel on screening CCTA.
* History of myocardial infarction (presumed type 1 event due to plaque rupture/erosion) and/or coronary revascularization by percutaneous coronary intervention.

Exclusion Criteria:

* History of coronary artery bypass graft (CABG).
* Moderate to severe renal dysfunction.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN), or total bilirubin (TBL) > 2 x ULN during screening.
* History of hemorrhagic stroke.
* History of major bleeding disorder.
* Planned cardiac surgery or arterial revascularization.
* Severe heart failure.
* Current, recent, or planned lipoprotein apheresis.
* Previously received ribonucleic acid therapy specifically targeting Lp(a).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2026-03-21 (Estimated); Primary Completion 2028-06-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Change in NCP Volume from Baseline to Week 72 | Baseline to Week 72

SECONDARY OUTCOMES:
Change in Low Attenuation Plaque Volume from Baseline to Week 72 | Baseline to Week 72
Change in Total Plaque Volume from Baseline to Week 72 | Baseline to Week 72
Change in Calcified Plaque Volume from Baseline to Week 72 | Baseline to Week 72
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 74

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com